CLINICAL TRIAL: NCT06689761
Title: Influence of Specific Collagen Peptides on Training-Induced Metabolic and Biomechanical Adaptations of Skeletal Muscle
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Collaborators: CRI Collagen Research Institute GmbH (Unknown)
Responsible Party: Principal Investigator, Kevin Bischof, Kevin Bischof Bakk., BSc., MSc., MBA, University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 01177
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Collagen Supplementation
Keywords: Running economy; collagen supplementation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ColCT (Experimental): Dietary Supplement: Collagen Participants ingest 15 grams specific collagen peptides daily
  + Concurrent training 12 weeks, 3x/week
  Interventions: Dietary Supplement: ColCT
- PlaCT (Placebo Comparator): Dietary Supplement: Placebo Participants ingest 15 grams of a placebo daily
  + Concurrent training 12 weeks, 3x/week
  Interventions: Dietary Supplement: PlaCT
- ColET (Experimental): Dietary Supplement: Collagen Participants ingest 15 grams specific collagen peptides daily
  + Endurance training 12 weeks, 3x/week
  Interventions: Dietary Supplement: ColET
- PlaET (Placebo Comparator): Dietary Supplement: Collagen Participants ingest 15 grams of placebo daily
  + Endurance training 12 weeks, 3x/week
  Interventions: Dietary Supplement: PlaET

INTERVENTIONS:
Dietary Supplement: ColCT — Dietary Supplement: Collagen Participants ingest 15 grams of specific collagen peptides daily
  Arms: ColCT
Dietary Supplement: ColET — Dietary Supplement: Collagen Participants ingest 15 grams of specific collagen peptides daily
  Arms: ColET
Dietary Supplement: PlaCT — Dietary Supplement: Placebo. Participants ingest 15 grams of placebo daily
  Arms: PlaCT
Dietary Supplement: PlaET — Dietary Supplement: Placebo. Participants ingest 15 grams of placebo daily
  Arms: PlaET

SUMMARY:
This study investigates whether taking daily collagen peptides, combined with long-term endurance or concurrent training can enhance running economy through muscle and/or tendon adaptations.

DETAILED DESCRIPTION:
An adequate and high-quality intake of proteins and amino acids is crucial for synthesizing the body's own connective tissue-like structures, such as muscles, tendons, ligaments, and bones. Various metabolic and hormonal processes are regulated or influenced by proteins. It is undisputed that measurable improvements are only possible through the combination of training and protein intake. Simply increasing protein intake without physical activity cannot be expected to result in structural or metabolic adaptations.

In recent years, interest in regular collagen intake in sports nutrition, particularly in connection with moderate to intense physical activity, has increased. Since collagen and its peptides are primarily found in force-transmitting structures such as tendons, studies have been conducted to examine how tendons adapt to collagen peptide supplementation. Studies by Jerger et al. (2022 & 2023) have shown that both the patellar and Achilles tendons adapt to collagen supplementation, as evidenced by an increased cross-sectional area compared to a non-caloric placebo. This increase allows tendons to withstand greater forces, making them more resilient and thus playing an important role in injury prevention. These results were achieved with a dose of 5g of collagen combined with three months of strength training.

Additionally, multi-month collagen peptide supplementation combined with concurrent training (strength and endurance training in one session) led to improved endurance performance. Both running distance and speed at the aerobic and anaerobic thresholds significantly increased compared to a placebo group with a daily intake of 15g of collagen over three months (Jerger et al. 2023, Jendricke et al. 2020).

Based on these results, the question arises as to whether regularly supplemented collagen peptides, combined with pure endurance training, lead to similar metabolic and/or tendon-specific adaptations. Therefore, the aim of this proposed study is to investigate both metabolic and specific (morphological, mechanical, and material) properties of the Achilles and patellar tendons to determine the mechanism through which the so-called "running economy" develops in connection with collagen peptides. The results will be compared to those of concurrent training, which has already shown metabolic adaptations as described above.

ELIGIBILITY:
Inclusion Criteria:

Male gender Age 18-40 years No subjective symptoms during physical exertion BMI of 18.5 to 26 Stable weight and dietary habits No extensive strength/endurance training (less than 3 hours per week) No contraindications to physical exertion according to ACSM guidelines No contraindications to supplemental nutrition or ergogenic supplements

Exclusion Criteria:

Contraindications to physical activity (e.g., chronic heart disease, arrhythmia, heart valve disease, arthritis, etc.; general exclusion criteria according to ACSM 2009; intolerance/aversion to animal protein) Arterial hypertension (systolic BP > 200 mmHg and/or diastolic BP > 105 mmHg) at rest Insulin-dependent diabetes mellitus (IDDM) Liver and/or kidney disease that excludes a high protein load

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — men
Enrollment: 60 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
One-hour time trial performance | Baseline and after 12 weeks
  Participants run an hour on the track outside as far as possible
Achilles tendon cross sectional-area | Baseline and after 12 weeks
  Ultrasound
Achilles and Patellar tendon Stiffness | Baseline and after 12 weeks
  Ultrasound + isokinetic dynamometer
VO2max | Baseline and after 12 weeks
  treadmill with spirometry

SECONDARY OUTCOMES:
Body composition | Baseline and after 12 weeks
  Fat mass, fat-free mass, extracellular mass, body cell mass, skeletal muscle mass. Measured by bioelectrical impedance analysis
Achilles tendon stress, strain, Young's modulus | Baseline and after 12 weeks
  Ultrasound + isokinetic dynamometer
Patellar tendon strain | Baseline and after 12 weeks
  Ultrasound + isokinetic dynamometer
RER, VT1, VT2, LTP1, LTP2, HFrel., FATox. | Baseline and after 12 weeks
  treadmill with spirometry and blood (lactate) collection.
Achilles tendon echointensity | Baseline and after 12 weeks
  Ultrasound

OTHER OUTCOMES:
Energy and macronutrient intake | Baseline and after 12 weeks
  kcal, protein, carbs, fat. 2x 3 day questionnaire (start and end of study)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Sport Science and University Sports, Department of Sport and Human Movement Science, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No